CLINICAL TRIAL: NCT03177083
Title: Open-label, Randomized, 2-arm, Active Comparator Study to Evaluate Safety and Tolerability in Portuguese Patients With Relapsing Remitting Multiple Sclerosis (MS) Transitioning From Current Subcutaneous Interferon Therapy to Peginterferon Beta 1a (PLEGRIDY™)
Brief Title: Evaluate Safety/Tolerability in Portuguese Participants With RRMS Transitioning From Current Therapy
Acronym: PLENO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRT-PEG-15-10880; 2016-000434-21 (EudraCT Number)
Record Dates: First submitted 2017-01-26; First posted 2017-06-06 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — peginterferon beta-1a; Interferon beta-1a; Interferon beta-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peginterferon beta-1a (Active Comparator)
  Interventions: Drug: peginterferon beta-1a
- Current Therapy (Active Comparator)
  Interventions: Drug: interferon beta-1a; Drug: interferon beta-1b

INTERVENTIONS:
Drug: peginterferon beta-1a — SC every 2 weeks
  Other Names: PLEGRIDY, BIIB017
  Arms: peginterferon beta-1a
Drug: interferon beta-1a — Per Summary of Product Characteristics (SMPC)
  Other Names: Rebif
  Arms: Current Therapy
Drug: interferon beta-1b — Per SMPC
  Other Names: Betaferon, Extavia
  Arms: Current Therapy

SUMMARY:
The primary objective of the study is to evaluate safety and tolerability as defined by the frequency of the adverse events (AEs) of flu-like symptoms (FLS) [chills, pyrexia, myalgia, and asthenia], injection site reactions (ISRs), and injection site reaction pain (ISR-P), over 24 weeks of treatment (the active comparator period) with PLEGRIDY 125 microgram (μg) subcutaneous (SC) every 2 weeks versus current SC IFN-β therapy in participants with Relapsing Remitting Multiple Sclerosis (RRMS).

ELIGIBILITY:
Key Inclusion Criteria:

* A confirmed diagnosis of RRMS, as defined by McDonald criteria (2017).
* An EDSS score between 0 and 5.0.
* All female participants of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 3 months after their last dose of study treatment.
* On continual treatment for ≥6 months with a single current SC IFN-β therapy, including IFN-β-1b 0.25 mg SC every other day or IFN-β-1a 22 μg or 44 μg SC 3 times weekly

Key Exclusion Criteria:

* Known history of human immunodeficiency virus.
* Known history of or positive test result for antibodies to hepatitis C, or current hepatitis B infection (defined as positive for hepatitis B surface antigen [HBsAg] and/or positive for hepatitis B core antibody [HBcAb]) at Screening. Participants with immunity to hepatitis B from either active vaccination (defined as negative HBsAg, positive hepatitis B surface antibody [HBsAb], and negative HBcAb) or from previous natural infection (defined as negative HBsAg, positive HBsAb immunoglobulin G, and positive HBcAb) are eligible to participate in the study (definitions are based on the Centers for Disease Control and Prevention's interpretation of the hepatitis B serology panel [CDC 2007]).
* An MS relapse that has occurred within the 50 days prior to randomization and/or lack of stabilization from a previous relapse prior to randomization (Day 1).
* Any previous treatment with PLEGRIDY.

NOTE: Other protocol defined Inclusion/Exclusion may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

PRIMARY OUTCOMES:
Combined Counts of Adverse Events (AEs) of Flu-Like Symptoms (FLS) | Up to Week 24
  FLS as defined by chills, pyrexia, myalgia, and asthenia
Combined Counts of AEs of Injection Site Reactions (ISRs) | Up to Week 24
  Defined as a post-application assessment score ≥2 in participant assessments using the Patient's Erythema Self-Assessment 1 (PSA) scale
Combined Counts of AEs of Injection Site Reactions (ISRs) | Up to Week 24
  Defined as a post-application assessment score ≥2 in clinician assessments using the Clinician Erythema Assessment (CEA) scale
Combined Counts of AEs of ISR Pain (ISRP) | Up to Week 24
  Defined as visual analog scale (VAS) associated with ISR ≥1 immediately after injection or 30 minutes post-injection

SECONDARY OUTCOMES:
Change in Participant-Reported Treatment Satisfaction Using Treatment Satisfaction Questionnaire for Medication (TSQM-9) in Participants Treated with PLEGRIDY Versus Current SC IFN-β | Baseline to Week 24
  A questionnaire assessing patient satisfaction with drug on 3 scales: effectiveness, convenience, and global satisfaction
Change in Participant-Reported Treatment Satisfaction Using TSQM-9 in Participants Who Switched from Current SC IFN-Β Therapy to PLEGRIDY at the End of the Comparator Period | Week 24 and Week 48
  A questionnaire assessing patient satisfaction with drug on 3 scales: effectiveness, convenience, and global satisfaction
Change in Participant-Reported Outcome (PRO) Measures in EuroQol Group 5-Dimension 3-Level Version (EQ-5D-3L) Index in Participants Treated with PLEGRIDY Versus Current SC IFN-Β | Baseline and Week 24
  The EQ-5D-3L is a standardized instrument for use as a measure of health outcome. It is a health questionnaire that consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems.
Change in PRO Measures in EQ-5D-3L Index in Participants Continuously Treated with PLEGRIDY Versus Participants Who Switched from Current SC IFN-Β Therapy to PLEGRIDY at the End of the Comparator Period | Week 24, Week 48 and Week 72
  The EQ-5D-3L is a standardized instrument for use as a measure of health outcome. It is a health questionnaire that consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems.
Change in PRO Measures in EQ-5D-3L Index in Participants Who Switched from Current SC IFN-Β Therapy to PLEGRIDY at the End of the Comparator Period | Baseline, Week 24, Week 48 and Week 72
  The EQ-5D-3L is a standardized instrument for use as a measure of health outcome. It is a health questionnaire that consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems.
Change in PRO Measures in Work Productivity and Activity Impairment Questionnaire: Multiple Sclerosis V2.1 (WPAI: MS) Score in Participants Treated with PLEGRIDY Versus Current SC IFN-Β | Baseline and Week 24
  The Work Productivity and Activity Impairment (WPAI) questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteesism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Change in PRO Measures in WPAI: MS Score in Participants Continuously Treated with PLEGRIDY Versus Participants Who Switched from Current SC IFN-Β Therapy to PLEGRIDY at the End of the Comparator Period | Week 24, Week 48 and Week 72
  The Work Productivity and Activity Impairment (WPAI) questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteesism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Change in PRO Measures in WPAI: MS Score in Participants Who Switched from Current SC IFN-Β Therapy to PLEGRIDY at the End of the Comparator Period | Baseline, Week 24, Week 48 and Week 72
  The Work Productivity and Activity Impairment (WPAI) questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteesism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity.
Percentage of Participants with Changes in Clinical Status Assessed Using the Expanded Disability Status Scale (EDSS) | Week 48
  The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist.
Change in PRO Measures in 12-Item Short Form Survey (SF-12) Score in Participants Treated with PLEGRIDY Versus Current SC IFN-Β | Baseline and Week 24
  A short form survey with 12 questions selected from the SF-36 Health Survey. The questions are weighted and summed to create two scales on physical and mental functioning. Physical Composite Scores (PCS) and Mental Composite Scores (MCS) range from 0 to 100, where a zero indicates the lowest level of health and 100 indicates the highest level of health.
Change in PRO Measures in SF-12 Score in Participants Continuously Treated with PLEGRIDY Versus Participants Who Switched from Current SC IFN-Β Therapy to PLEGRIDY at the End of the Comparator Period | Week 24, Week 48 and Week 72
  A short form survey with 12 questions selected from the SF-36 Health Survey. The questions are weighted and summed to create two scales on physical and mental functioning. Physical Composite Scores (PCS) and Mental Composite Scores (MCS) range from 0 to 100, where a zero indicates the lowest level of health and 100 indicates the highest level of health.
Change in PRO Measures in SF-12 Score in Participants Who Switched from Current SC IFN-Β Therapy to PLEGRIDY at the End of the Comparator Period | Baseline, Week 24, Week 48 and Week 72
  A short form survey with 12 questions selected from the SF-36 Health Survey. The questions are weighted and summed to create two scales on physical and mental functioning. Physical Composite Scores (PCS) and Mental Composite Scores (MCS) range from 0 to 100, where a zero indicates the lowest level of health and 100 indicates the highest level of health.
Change in PRO Measures in Fatigue Severity Scale (FSS) Score in Participants Treated with PLEGRIDY Versus Current SC IFN-Β | Baseline and Week 24
  A 9-item questionnaire that measures the severity of fatigue and functionality. Each question is scored on a scale of 1 to 7, where 1 equals strongly disagree and 7 equals strongly agree. A higher total score indicates greater fatigue severity and impairment.
Change in PRO Measures in FSS Score in Participants Continuously Treated with PLEGRIDY Versus Participants Who Switched from Current SC IFN-Β Therapy to PLEGRIDY at the End of the Comparator Period | Week 24, Week 48 and Week 72
  A 9-item questionnaire that measures the severity of fatigue and functionality. Each question is scored on a scale of 1 to 7, where 1 equals strongly disagree and 7 equals strongly agree. A higher total score indicates greater fatigue severity and impairment.
Change in PRO Measures in FSS Score in Participants Who Switched from Current SC IFN-Β Therapy to PLEGRIDY at the End of the Comparator Period | Baseline, Week 24, Week 48 and Week 72
  A 9-item questionnaire that measures the severity of fatigue and functionality. Each question is scored on a scale of 1 to 7, where 1 equals strongly disagree and 7 equals strongly agree. A higher total score indicates greater fatigue severity and impairment.
Change in PRO Measures in Hospital Anxiety And Depression Scale (HADS) Score in Participants Treated with PLEGRIDY Versus Current SC IFN-Β | Baseline and Week 24
  A 14-item self-rating scale that assesses anxiety and depression. Each question is scored on a scale ranging from 0 to 3. Responses are summed to provide separate scores for anxiety and depression that range from 0 to 21. For each corresponding subscale, a total score of 0-7 equals normal, 8-10 equals borderline case, and 11-21 equals case.
Change in PRO Measures in HADS Score in Participants Continuously Treated with PLEGRIDY Versus Participants Who Switched from Current SC IFN-Β Therapy to PLEGRIDY at the End of the Comparator Period | Week 24, Week 48 and Week 72
  A 14-item self-rating scale that assesses anxiety and depression. Each question is scored on a scale ranging from 0 to 3. Responses are summed to provide separate scores for anxiety and depression that range from 0 to 21. For each corresponding subscale, a total score of 0-7 equals normal, 8-10 equals borderline case, and 11-21 equals case.
Change in PRO Measures in HADS Score in Participants Who Switched from Current SC IFN-Β Therapy to PLEGRIDY at the End of the Comparator Period | Baseline, Week 24, Week 48 and Week 72
  A 14-item self-rating scale that assesses anxiety and depression. Each question is scored on a scale ranging from 0 to 3. Responses are summed to provide separate scores for anxiety and depression that range from 0 to 21. For each corresponding subscale, a total score of 0-7 equals normal, 8-10 equals borderline case, and 11-21 equals case.
Participants Adherence to Study Treatment as Measured by Treatment Adherence Questionnaire | Week 24 and Week 72
  A questionnaire assessing adherence and the reasons for not taking drug at the recommended frequency of administration.
Participants Adherence to Study Treatment as Measured by Returned Injection Pens | Week 24 and Week 72
  Treatment adherence surveillance
Participants Adherence to Study Treatment as Measured by Treatment Adherence Questionnaire in Participants Who Switched from Current SC IFN-Β Therapy to PLEGRIDY at the End of the Comparator Period | Baseline, Week 24, Week 48 and Week 72
  A questionnaire assessing adherence and the reasons for not taking drug at the recommended frequency of administration.
Participants Adherence to Study Treatment as Measured by Returned Injection Pens in Participants Who Switched from Current SC IFN-Β Therapy to PLEGRIDY at the End of the Comparator Period | Baseline, Week 24, Week 48 and Week 72
  Treatment adherence surveillance
Proportion of Pain-Free Participants Immediately After Injection (Defined as 0 mm for All Full-Dose Injections on VAS of Participant-Reported Pain) at End Of the Comparator Period in Participants Treated with PLEGRIDY Versus Current SC IFN-Β | Week 24
  0 mm for all full-dose injections on Visual Analog Scale (VAS) of participant-reported pain.
Proportion of Pain-Free Participants 30 Minutes after Injection (Defined as 0 mm for All Full-Dose Injections on VAS of Participant-Reported Pain) at End of the Comparator Period in Participants Treated with PLEGRIDY Versus Current SC IFN-Β | Week 24
  0 mm for all full-dose injections on (VAS) of participant-reported pain.
Average Change in Participant-Reported VAS Pain Score from Pre-Injection to 30 Minutes Post-Injection in Participants Treated with PLEGRIDY Versus Current SC IFN-Β | Week 24
  Measured by participant-reported VAS pain score
Average Change in Participant-Reported VAS Pain Score from Pre-Injection to Immediate Post-Injection in Participants Treated with PLEGRIDY Versus Current SC IFN-Β | Week 24
  Measured by participant-reported VAS pain score
Percentage of Participants with Changes in Relapse Activity | Week 72
  Measured by change of ARR pre-study to on-study ARR
Annualized Relapse Rate (ARR) in Participants in the Overall Population | Week 72
  Calculated by dividing the total number of participant relapses by the total number of participant years at risk.
Proportion of Relapsed Participants in Overall Population | Week 72
  Proportion of total study participants who experienced a confirmed clinical relapse during the study.
Percentage of Participants with an Adverse Event (AE), Serious AE, and Discontinuations of Study Treatment due to an AE in Participants Treated with PLEGRIDY Versus Current SC IFN-β | Week 24
  Safety surveillance
Percentage of Participants with an AE, Serious AE, and Discontinuation of Study Treatment due to an AE Continuously Treated with PLEGRIDY | Week 24, Week 48 and Week 72
  Safety surveillance
Percentage of Participants with an AE, Serious AE, and Discontinuation of Study Treatment due to an AE Who Switched from Current SC IFN-Β Therapy to PLEGRIDY at the End of the Comparator Period | Week 24, Week 48 and Week 72
  Safety surveillance

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (15):
- Portugal (15):
  - Hospital Fernando Fonseca, Amadora
  - Hospital de Braga, Braga
  - Centro Hospitalar Cova da Beira, Covilha
  - Hospital Evora, Evora
  - Hospital Dr. Nelio Mendonça, Funchal
  - Hospital da Senhora da Oliveira, Guimarães
  - Centro Hospitalar de Leiria, Leiria
  - Hospital Egas Moniz, Lisbon
  - Hospital da Luz, Lisbon
  - Centro Hospitalar Lisboa Norte - Hosp Santa Maria, Lisbon
  - Hospital Beatriz Ângelo, EPE, Loures
  - ULS Matosinhos, Matosinhos Municipality
  - Hospital Santo Antonio, Porto
  - Hospital de Sao Sebastiao, Santa Maria da Feira
  - Hospital Viana do Castelo, Viana do Castelo